CLINICAL TRIAL: NCT00394732
Title: Effect of Lumbar Disc Prosthesis Versus Multidisciplinary Rehabilitation Program in Patients With Chronic Low Back Pain and Degenerative Disc. A Prospective Randomized Clinical Multicentre Trial.
Brief Title: Disc Prosthesis Versus Multidisciplinary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); St. Olavs Hospital (Other); University of Tromso (Other); Haukeland University Hospital, Dept of neck and back diseases (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); Falu Lasarett Röntgen (Other)
Responsible Party: Principal Investigator, Kjersti Storheim, PhD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201006
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Low Back Pain; Degenerative Disc Disease
Keywords: chronic low back pain; total disc replacement; multidisciplinary rehabilitation; clinical effects; cost effectiveness; randomized controlled trial; multicenter study
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Device: Total Disc Prosthesis
Behavioral: Multidisciplinary rehabilitation program

SUMMARY:
Surgical methods offered to patients with chronic low back pain are controversial. In addition, new and expensive treatment methods like total disc replacemet (TDR) are a challenge for the health care services. At present, ongoing randomized studies in both Europe and USA are comparing TDR to fusion. However, to our knowledge, no randomized trials have compared TDR to non-surgical treatment. The aim of the present study is to evaluate the effect of a comprehensive and structured non-surgical treatment with TDR surgery in patients with chronic low back pain and localized degenerative disc changes.

Main hypothesis: There is no difference in treatment effect between surgery with lumbar total disc prosthesis and a multidisciplinary rehabilitation program measured by Oswestry Disability Index after 1 and 2 years.

Secondary hypothesis: There is no difference in cost - effectiveness between surgery with lumbar disc prosthesis and a multidisciplinary rehabilitation program after 1 and 2 years.

DETAILED DESCRIPTION:
Description of interventions.

Surgical intervention: The surgical intervention consists of replacement of the degenerative intervertebral lumbar disc with a artificial lumbar disc device (ProDisc II, Spine Solutions Inc. , New York, NY). The ProDisc consists of three pieces, two metal endplates and a polyethylene core that is fixed to the inferior endplate when the device is implanted, and is implanted through a retroperitoneal (or transperitoneal) access. Depending on the surgeon, a Pfannenstiel incision or a para median incision is used. A fluoroscope is used to ensure that the prosthesis is placed in the midline and sufficiently towards the posterior edge of the corpus vertebrae. All hospitals participating in the study will use the same artificial lumbar disc device, and standard instruments from the manufacturer are used for inserting the disc. Postoperatively, orthoses will not be used, but patients are given restrictions on heavy lifting and excessive movements the first 6 weeks after surgery. Otherwise, no instructions will be given. Six weeks after surgery, patients will be referred to physiotherapy.

Non-surgical intervention: The intervention is based on a treatment model described by Brox et al (Spine 2003;28:1913-1921) and consists of a cognitive approach and supervised physical exercise. The treatment is interdisciplinary and is directed by a team of physiotherapists and specialists in physical medicine and rehabilitation. The intervention is organized as an outpatient treatment in groups of 6 - 8 patients during a period of 12 - 15 treatment days. In agreement with the patient, individual goals for the rehabilitation process are established.

Sub-studies:

Several sub - projects will be conducted at the different hospitals in the study, in example validation of discography, RSA to validate the migration and motion of the prosthesis, a biomechanical study using DCRA technique, validation of a classification system for physiotherapy and a responsiveness of questionnaires included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain as the main symptom for at least one year.
* Structured physiotherapy or chiropractic treatment for at least 6 months without (significant) effect.
* Oswestry Disability Index score of 30% points or more
* Degenerative changes in the intervertebral disc in one or both of the two lowest levels of the lumbar spine (L4/L5 and/or L5/S1). (Degenerative changes are classified based on MR findings according to the following criteria: At least 40% reduction of disc height, Modic changes type I and/or II, "High intensity zone" in the disc, Morphological changes classified as changes in signal intensity in the disc. To classify the disc as degenerative the first criteria alone or at least two of the other criteria must be present. The MR series are evaluated by two independent observers.)

Exclusion Criteria:

* Generalized chronic pain syndrome (widespread myofascial pain)
* Degeneration established in more than two levels. To be classified as a normal disc, the disc height must not be reduced more than 40% and all other criteria of degenerative disc disease aforementioned must be absent. The classification of a normal disc is performed by two independent observers. If disagreement, the pictures will be classified by a third observer and the outcome decided by simple majority.
* Symptoms of spinal stenosis
* Disc protrusion or recess stenosis with nerve root affection
* Spondylolysis
* Isthmic spondylolisthesis
* Arthritis
* Former fracture of L1 - S1
* Ongoing psychiatric or somatic disease that excludes either one or both treatment alternatives
* Does not understand Norwegian language, spoken or in writing
* Drug abuse
* Osteoporosis
* Congenital or acquired deformity

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2004-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index
Cost-effectiveness (full economic analysis)

SECONDARY OUTCOMES:
Side effects
Time out of work
Fear - avoidance beliefs
Self - efficacy for pain
Hopkins symptoms check list
Drug consumption
Life satisfaction (EQ 5D and SF - 36)
Pain (low back pain and leg pain) on VAS

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Storheim, PT, PhD, Study Director — Orthopedic Centre, Ullevål University Hospital / NAR
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen, Bergen
  - Ullevål University Hospital, Orthopedic Centre, Oslo, Oslo County
  - Stavanger University Hospital, Stavanger, Stavanger
  - University Hospital of Nothern-Norway, Tromsø, Tromsø
  - St.Olavs Hospital, NSSL, Trondheim, Trondheim

REFERENCES:
- [Result] Hellum C, Johnsen LG, Storheim K, Nygaard OP, Brox JI, Rossvoll I, Ro M, Sandvik L, Grundnes O; Norwegian Spine Study Group. Surgery with disc prosthesis versus rehabilitation in patients with low back pain and degenerative disc: two year follow-up of randomised study. BMJ. 2011 May 19;342:d2786. doi: 10.1136/bmj.d2786. PMID 21596740
- [Result] Hellum C, Berg L, Gjertsen O, Johnsen LG, Neckelmann G, Storheim K, Keller A, Grundnes O, Espeland A; Norwegian Spine Study Group. Adjacent level degeneration and facet arthropathy after disc prosthesis surgery or rehabilitation in patients with chronic low back pain and degenerative disc: second report of a randomized study. Spine (Phila Pa 1976). 2012 Dec 1;37(25):2063-73. doi: 10.1097/BRS.0b013e318263cc46. PMID 22706091
- [Result] Hellum C, Johnsen LG, Gjertsen O, Berg L, Neckelmann G, Grundnes O, Rossvoll I, Skouen JS, Brox JI, Storheim K; Norwegian Spine Study Group. Predictors of outcome after surgery with disc prosthesis and rehabilitation in patients with chronic low back pain and degenerative disc: 2-year follow-up. Eur Spine J. 2012 Apr;21(4):681-90. doi: 10.1007/s00586-011-2145-3. Epub 2012 Jan 13. PMID 22246644
- [Derived] Storheim K, Berg L, Hellum C, Gjertsen O, Neckelmann G, Espeland A, Keller A; Norwegian Spine Study Group. Fat in the lumbar multifidus muscles - predictive value and change following disc prosthesis surgery and multidisciplinary rehabilitation in patients with chronic low back pain and degenerative disc: 2-year follow-up of a randomized trial. BMC Musculoskelet Disord. 2017 Apr 4;18(1):145. doi: 10.1186/s12891-017-1505-5. PMID 28376754
- [Derived] Johnsen LG, Brinckmann P, Hellum C, Rossvoll I, Leivseth G. Segmental mobility, disc height and patient-reported outcomes after surgery for degenerative disc disease: a prospective randomised trial comparing disc replacement and multidisciplinary rehabilitation. Bone Joint J. 2013 Jan;95-B(1):81-9. doi: 10.1302/0301-620X.95B1.29829. PMID 23307678